CLINICAL TRIAL: NCT01926743
Title: Identification of Complete Lymph Node Removal by Application of Near Infrared Fluorescence Imaging in Laparoscopic and Robotic Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2013-0414
Record Dates: First submitted 2013-08-18; First posted 2013-08-21 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Gastric Cancer
Keywords: near infrared; fluorescence imaging; indocyanine green; gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NIR with ICG group (Experimental)
  Interventions: Procedure: Near infrared fluorescence imaging during laparoscopic or robotic gastrectomy

INTERVENTIONS:
Procedure: Near infrared fluorescence imaging during laparoscopic or robotic gastrectomy — 0.75mg of ICG injection around tumor each four direction by endoscopy on one or two days before surgery. NIR fluorescence imaging application during laparoscopic or robotic gastrectomy

SUMMARY:
Lymph node dissection in gastric cancer surgery is a very important factor not only for exact acquisition of stage but also proper treatment. Realistically, it is impossible to identify complete removal of lymph node in dissected nodal station by naked eye. The investigators can assess the route of lymphatic drainage and identify residual lymph nodes in dissected area. In the field of gastric cancer treatment, ICG and near infra-red fluorescence imaging was used only detection of sentinel lymph nodes. However, this novel concept can help to understand lymphatic drainage and make surgeons to perform D1+ or D2 lymph node dissection completely.

ELIGIBILITY:
Inclusion Criteria:

1. Males or Females, aged≥20 years and ≤80 years
2. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 or 1 at study entry
3. American Society of Anesthesiolosists (ASA) score of 1 to 3
4. Histologically confirmed adenocarcinoma in stomach
5. Clinical stage I (T1N0M0, T2N0M0, T1N1M0)

5. The patient has curatively resectable disease 6. The patient has given their written informed consent to participate in the study

Exclusion Criteria:

1. M1 status
2. Experience of previous gastric resection
3. Complication due to gastric cancer, such as complete obstruction or perforation
4. History of anti-cancer therapy (chemotherapy or radiotherapy) for current gastric cancer
5. History of surgery, chemotherapy or radiotherapy for primary carcinoma of other organ in 5 years

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2014-01-31 (Actual); Study Completion 2014-01-31 (Actual)

PRIMARY OUTCOMES:
To compare the number of retrieved lymph node in each nodal station after additional application of near infra-red fluorescence imaging | About 7 days after operation when pathologic result was reported

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Yonsei University Health System, Yonsei University College of Medicine, Seoul, South Korea

REFERENCES:
- [Background] Marano A, Priora F, Lenti LM, Ravazzoni F, Quarati R, Spinoglio G. Application of fluorescence in robotic general surgery: review of the literature and state of the art. World J Surg. 2013 Dec;37(12):2800-11. doi: 10.1007/s00268-013-2066-x. PMID 23645129
- [Background] Schaafsma BE, Mieog JS, Hutteman M, van der Vorst JR, Kuppen PJ, Lowik CW, Frangioni JV, van de Velde CJ, Vahrmeijer AL. The clinical use of indocyanine green as a near-infrared fluorescent contrast agent for image-guided oncologic surgery. J Surg Oncol. 2011 Sep 1;104(3):323-32. doi: 10.1002/jso.21943. Epub 2011 Apr 14. PMID 21495033
- [Background] Rossi EC, Ivanova A, Boggess JF. Robotically assisted fluorescence-guided lymph node mapping with ICG for gynecologic malignancies: a feasibility study. Gynecol Oncol. 2012 Jan;124(1):78-82. doi: 10.1016/j.ygyno.2011.09.025. Epub 2011 Oct 11. PMID 21996262
- [Background] Ohdaira H, Nimura H, Fujita T, Mitsumori N, Takahashi N, Kashiwagi H, Narimiya N, Yanaga K. Tailoring treatment for early gastric cancer after endoscopic resection using sentinel node navigation with infrared ray electronic endoscopy combined with indocyanine green injection. Dig Surg. 2009;26(4):276-81. doi: 10.1159/000227766. Epub 2009 Jul 8. PMID 19590206
- [Background] Nimura H, Narimiya N, Mitsumori N, Yamazaki Y, Yanaga K, Urashima M. Infrared ray electronic endoscopy combined with indocyanine green injection for detection of sentinel nodes of patients with gastric cancer. Br J Surg. 2004 May;91(5):575-9. doi: 10.1002/bjs.4470. PMID 15122608
- [Background] Koyama T, Tsubota A, Nariai K, Mitsunaga M, Yanaga K, Takahashi H. Novel biomedical imaging approach for detection of sentinel nodes in an experimental model of gastric cancer. Br J Surg. 2007 Aug;94(8):996-1001. doi: 10.1002/bjs.5650. PMID 17380563
- [Background] Jeschke S, Lusuardi L, Myatt A, Hruby S, Pirich C, Janetschek G. Visualisation of the lymph node pathway in real time by laparoscopic radioisotope- and fluorescence-guided sentinel lymph node dissection in prostate cancer staging. Urology. 2012 Nov;80(5):1080-6. doi: 10.1016/j.urology.2012.05.050. Epub 2012 Sep 15. PMID 22990053
- [Background] Cahill RA, Anderson M, Wang LM, Lindsey I, Cunningham C, Mortensen NJ. Near-infrared (NIR) laparoscopy for intraoperative lymphatic road-mapping and sentinel node identification during definitive surgical resection of early-stage colorectal neoplasia. Surg Endosc. 2012 Jan;26(1):197-204. doi: 10.1007/s00464-011-1854-3. Epub 2011 Aug 19. PMID 21853392